CLINICAL TRIAL: NCT05516953
Title: Clinical Study Evaluating the Efficacy of Baclofen in Preventing Postoperative Nausea and Vomiting After Laparoscopic Sleeve Gastrectomy
Brief Title: Baclofen in Preventing Postoperative Nausea and Vomiting After Bariatric Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Gamal Moussa, Assistant Lecturer at Clinical Pharmacy department , Faculty of Pharmacy -Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 35647/8/22
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Nausea and Vomiting; Laparoscopic Sleeve Gastrectomy; Morbid Obesity
Keywords: Postoperative Nausea and Vomiting; Laparoscopic Sleeve Gastrectomy; baclofen; Morbid Obesity
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Obesity, Morbid | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1(Control group) (No Intervention): include 50 patients scheduled for sleeve gastrectomy
- Group 2 (Experimental): which include 50 patients scheduled for sleeve gastrectomy
  Interventions: Drug: Baclofen Tablets

INTERVENTIONS:
Drug: Baclofen Tablets — 10 mg oral baclofen 1 h before anesthesia
  Other Names: baclofen
  Arms: Group 2

SUMMARY:
This study aims to evaluate the possible efficacy of baclofen on postoperative nausea and vomiting in patient with morbid obesity who will undergo laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
. A total of 100 morbidly obese patients who will be scheduled for sleeve gastrectomy will be included in the study. The patients will be selected from those attending Gastrointestinal and Laparoscopic Surgery Unit, General Surgery Department, Tanta University Hospital, Tanta, Egypt. The participants will be randomized into four groups by closed envelop method

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients scheduled for sleeve gastrectomy with BMI ≥35 kg/m2 with the presence of comorbidity such as hypertension, arthritis, and diabetes.
* Morbidly obese patients scheduled for sleeve gastrectomy with BMI ≥ 40 kg/m2 without comorbidity.
* Patients fit for anesthesia and surgery.

Exclusion Criteria:

* Patients with BMI >55 kg/m2.
* Patients with previous procedures for the treatment of obesity.
* Pregnant females and lactating women.
* Patients with psychological or psychiatric disease
* Administration of antiemetic medication or systemic corticosteroids within 24 hours before surgery
* Patients who experienced vomiting within 24 hours before surgery.
* Patients with history of alcohol or drug abuse.
* Patients with hypersensitivity or contraindications to any of the drugs used in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study will be the complete response | The first 48 hours after surgery.
  Complete response is defined as the absence of PONV and the lack of a need for rescue antiemetic therapy.

SECONDARY OUTCOMES:
Change in serum level of vasopressin | The first 48 hours after surgery.
  Blood samples will be collected at baseline, 24 hours and 48 hours after surgery
Change in serum level of substance P | The first 48 hours after surgery.
  Blood samples will be collected at baseline, 24 hours and 48 hours after surgery
Change in serum level of dopamine | The first 48 hours after surgery.
  Blood samples will be collected at baseline, 24 hours and 48 hours after surgery
Change in serum level of serotonin | The first 48 hours after surgery.
  Blood samples will be collected at baseline, 24 hours and 48 hours after surgery
Change in serum level of tachykinin 1 | The first 48 hours after surgery.
  Blood samples will be collected at baseline, 24 hours and 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aya Moussa, Principal Investigator — Tanta University
Locations (1):
- Gastrointestinal and Laparoscopic Surgery Unit, General Surgery Department, Tanta University Hospital., Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No